CLINICAL TRIAL: NCT05855993
Title: Effects of Neural Glides With and Without Therapeutic Ultra Sound on Pain Symptom Severity and Functional Status in Pregnant Computer Workers With Carpal Tunnel Syndrome
Brief Title: Neural Glides With and Without Therapeutic Ultra Sound on in Pregnant Computer Workers With Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0520
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy Related
Keywords: CTS; Functional Status Scale; Non Invasive Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve Glide Exercise with Ultra Sound (Experimental)
  Interventions: Other: Nerve Glide Exercise with Ultra Sound
- Nerve Glide Exercise without Ultra Sound (Active Comparator)
  Interventions: Other: Nerve Glide Exercise without Ultra Sound

INTERVENTIONS:
Other: Nerve Glide Exercise with Ultra Sound — A brief demonstration will be given to perform the nerve glides exercises to both group. The duration of exercise programmed is 15 minutes every 3 to 5 times per day for 4 weeks. Group A will perform exercise with ultrasound
  Arms: Nerve Glide Exercise with Ultra Sound
Other: Nerve Glide Exercise without Ultra Sound — Group B will perform exercise for 10 minutes every 3 to 5 times per day without ultrasound.
  Arms: Nerve Glide Exercise without Ultra Sound

SUMMARY:
To study the effects of Neural Glides with and without using therapeutic ultrasound and functional status in pregnant computer workers with CTS

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome is a median nerve compression and results in significant discomfort and pain, daily living activity limitation, loss of sleep and work disability. Carpal tunnel Syndrome is more common in pregnancy because in pregnancy prolactin hormone increase the fluid retention in extra capsule and results in soft tissue swelling. Several therapeutically treatments have been advocated for the carpal tunnel syndrome including Mobilizations, nerve gliding, tendon gliding, Ultrasound, icing, Massaging. Women experience pregnancy several times, and if they acquire Carpal tunnel syndrome, invasive treatments cannot be used, the probability of reoccurrence of Carpal tunnel syndrome in the next pregnancy with higher intensity. Use of non-invasive treatment methods are more beneficial. Carpal tunnel syndrome very common nowadays as most of the population is involved in computer work by some means especially the computer working ladies who always use the conventional mouse and key board for their work. Pregnant Women diagnosed with Carpal Tunnel syndrome and are computer working would be selected for this study. Diagnostic criteria would be positive Tinel's and Phalen's. The subjects will be divided into two groups. Group A (Experimental) and group B (Control). Group A will perform with nerve glides with therapeutic ultrasound. The control group does only exercise program (tendon and nerve gliding exercises). Both groups are assessed by outcome measures pre and post interventions. Pain symptoms is measured with the help of Visual Analogue Scale, The Boston Carpal Tunnel questionnaire form will administer for the patient evaluation Functional Status Scale and Symptom Severity Scale.

ELIGIBILITY:
Inclusion Criteria:

Third trimester Tinel's sign positive Phalen test positive Pregnant women with pain and numbness in wrist and fingers Women with tingling sensation in the wrist Nocturnal parasthesia in wrist and fingers

Exclusion Criteria:

Inflammatory joint disease Age above 35 years Wrist bone fractures Hand surgery Diabetes Gout Autoimmune disease Person with rheumatoid arthritis Any other abnormalities

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | 4 Week
  To calculate score, add together the scores for all 11 questions in part 1, to give a total out of 55.(11)

SECONDARY OUTCOMES:
Visual Analog Scale(VAS) | 4 weeks
  To measure the pain response before and after treatment as no pain (0)severe pain (10)

OTHER OUTCOMES:
Symptom Severity Scale (SSS) | 4 weeks
  Measure the severity of symptom. Scores mild, moderat, severe & very severe
Functional Status Scale (FSS) | 4 weeks
  Used to measure the functional disability of hand. Scoring - No difficulty, mild difficulty, moderate difficulty & cant do at all

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Mahjabeen, PhD, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashour AA, Yehia RM, ElMeligie MM, Hanafy AF. Effectiveness of high intensity laser therapy on pain, grip strength and median nerve conductivity in pregnant women with carpal tunnel syndrome: A randomized controlled trial. J Hand Ther. 2023 Jul-Sep;36(3):536-545. doi: 10.1016/j.jht.2022.03.005. Epub 2022 Jul 8. PMID 35817691
- [Background] Oliveira GAD, Bernardes JM, Santos ES, Dias A. Carpal tunnel syndrome during the third trimester of pregnancy: prevalence and risk factors. Arch Gynecol Obstet. 2019 Sep;300(3):623-631. doi: 10.1007/s00404-019-05233-6. Epub 2019 Jul 2. PMID 31267198
- [Background] Keskin Y, Kilic G, Taspinar O, Posul SO, Halac G, Eren F, Erol E, Urkmez B, Aydin T. Effectiveness of home exercise in pregnant women with carpal tunnel syndrome: Randomized Control Trial. J Pak Med Assoc. 2020 Feb;70(2):202-207. doi: 10.5455/JPMA.1846. PMID 32063607
- [Background] Bartkowiak Z, Eliks M, Zgorzalewicz-Stachowiak M, Romanowski L. The Effects of Nerve and Tendon Gliding Exercises Combined with Low-level Laser or Ultrasound Therapy in Carpal Tunnel Syndrome. Indian J Orthop. 2019 Mar-Apr;53(2):347-352. doi: 10.4103/ortho.IJOrtho_45_17. PMID 30967707
- [Background] Nageswari C, Meena N, Devi TR. A Non Invasive Approach to Prevent Carpel Tunnel Syndrome of IT Women during Pregnancy
- [Background] VAIDYA S, NARIYA D. Effect of Neural Mobilisation Versus Nerve and Tendon Gliding Exercises in Carpal Tunnel Syndrome: A Randomised Clinical Trial. Journal of Clinical & Diagnostic Research. 2020;14(6)
- [Background] Sim SE, Gunasagaran J, Goh KJ, Ahmad TS. Short-term clinical outcome of orthosis alone vs combination of orthosis, nerve, and tendon gliding exercises and ultrasound therapy for treatment of carpal tunnel syndrome. J Hand Ther. 2019 Oct-Dec;32(4):411-416. doi: 10.1016/j.jht.2018.01.004. Epub 2018 Feb 13. PMID 29426574
- [Background] Wolny T, Saulicz E, Linek P, Shacklock M, Mysliwiec A. Efficacy of Manual Therapy Including Neurodynamic Techniques for the Treatment of Carpal Tunnel Syndrome: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2017 May;40(4):263-272. doi: 10.1016/j.jmpt.2017.02.004. Epub 2017 Apr 8. PMID 28395984
- [Background] Kadam P, Bhalerao S. Sample size calculation. Int J Ayurveda Res. 2010 Jan;1(1):55-7. doi: 10.4103/0974-7788.59946. No abstract available. PMID 20532100
- [Background] Price DD, Staud R, Robinson ME. How should we use the visual analogue scale (VAS) in rehabilitation outcomes? II: Visual analogue scales as ratio scales: an alternative to the view of Kersten et al. J Rehabil Med. 2012 Sep;44(9):800-1; discussion 803-4. doi: 10.2340/16501977-1031. No abstract available. PMID 22915047
- [Background] Bougea A, Zambelis T, Voskou P, Katsika PZ, Tzavara C, Kokotis P, Karandreas N. Reliability and Validation of the Greek Version of the Boston Carpal Tunnel Questionnaire. Hand (N Y). 2018 Sep;13(5):593-599. doi: 10.1177/1558944717725379. Epub 2017 Aug 20. PMID 28825339